CLINICAL TRIAL: NCT00050596
Title: A Randomized Study Comparing 4 Monthly Doses of MDX-010 (CTLA-4) as a Single Agent or Used in Combination With a Single Dose of Docetaxel in Patients With Hormone-Refractory Prostate Cancer
Brief Title: Comparison Study of MDX-010 (CTLA-4) Alone and Combined With Docetaxel in the Treatment of Patients With Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MDX010-07; CA184-019 (Other: BMS)
Record Dates: First submitted 2002-12-16; First posted 2002-12-17 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ipilimumab; Docetaxel

INTERVENTIONS:
Drug: MDX-010 / MDX-010 + Docetaxel

SUMMARY:
The primary objectives of the study are to determine the safety and activity of multiple doses of MDX-010 in patients with hormone-refractory prostate cancer (HRPC), and to determine the safety and activity profile of a single dose of cytotoxic chemotherapy (docetaxel) in combination with MDX-010

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of adenocarcinoma of the prostate.
* Metastatic prostate cancer (positive bone scan or measurable disease).
* Progressive disease after androgen deprivation.
* No prior chemotherapy or immunotherapy (tumor vaccine, cytokine, or growth factor given to control prostate cancer).

Exclusion Criteria:

* Other prior malignancy, except for adequately treated basal or squamous cell skin cancer or superficial bladder cancer, or any other cancer from which the patient has been disease-free for greater than or equal to 5 years.
* Previous occurrence of autoimmune disease.
* Active infection requiring therapy including HIV or chronic hepatitis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-11; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (11):
- United States (11):
  - Advanced Clinical Therapeutics, Tucson, Arizona
  - Pacific Shores Medical Group, Long Beach, California
  - San Diego Uro-Research, San Diego, California
  - LSU Health Science Center/ Stanley S. Scott Cancer Center (uptown campus), New Orleans, Louisiana
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University Urological Research Institute, Providence, Rhode Island
  - Grand Strand Urology, Myrtle Beach, South Carolina
  - Urology Associates of North Texas, Arlington, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Salt Lake Research, Salt Lake City, Utah
  - Seattle Cancer Center Alliance, Seattle, Washington